CLINICAL TRIAL: NCT02692534
Title: Cocaine Use and General Anesthesia: A Prospective Study of Cardiovascular and Anesthetic Effects
Brief Title: Cocaine Use and Outcomes of General Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 062015-066
Record Dates: First submitted 2016-01-21; First posted 2016-02-26 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia
Keywords: Anesthesia; Cocaine Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cocaine negative: Patients with preoperative urine cocaine negative results
  Interventions: Other: Urine cocaine negative
- Cocaine positive: Patients with preoperative urine cocaine positive results
  Interventions: Other: Urine cocaine positive

INTERVENTIONS:
Other: Urine cocaine negative — Preoperative urine cocaine negative
  Groups: Cocaine negative
Other: Urine cocaine positive — Preoperative urine cocaine positive
  Groups: Cocaine positive

SUMMARY:
In this prospective study, investigators plan to evaluate the outcome of general anesthesia in the context of patients with a positive cocaine urine test. Patients with a positive urine cocaine test who do not appear acutely toxic and have normal vital signs may not have an increased rate of perioperative complications during elective surgery compared to similar patients with negative urine cocaine screening tests. Patients who are chronic cocaine users may have a higher anesthetic requirement.

DETAILED DESCRIPTION:
Patients with a history of cocaine abuse who are scheduled to undergo surgery at Parkland Hospital will be asked to provide a urine sample for a screening toxicology test on the day of surgery. Patients will also be asked to fill out a questionnaire with questions pertaining to their drug use history. The remaining aspects of perioperative care, including the general anesthetic technique, will be standardized for all patients and will not differ from the standard of care. The anesthesia faculty, resident, or CRNA will identify patients and obtain consent and ask the patient to fill out the questionnaire. This prospective study is intended to enroll about 300 cocaine positive and negative patients over a 2 year period.

Blood samples will be collected for analysis of cardiac troponin T (cTnT) pre- and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* ASA physical status classification 1 to 3
* Personal history of cocaine abuse
* Scheduled for a non-emergent operation that requires general anesthesia
* Vital signs within generally accepted ranges for normal [HR 60-100, RR 12-20, SpO2 > 96% on room air, BP 90-140/60-90 unless a diagnosis of hypertension is present, T 36-38 degrees)
* Willing and able to consent in English or Spanish

Exclusion Criteria:

* Age less than 18 or older than 70
* Unable to give informed consent for participation in the study
* Patient refusal
* Monitored anesthesia care (MAC) or regional anesthesia planned
* Pregnant or lactating
* Emergent surgery
* Acute cocaine intoxication based on clinical symptomatology (hypertension, tachycardia, agitation, delirium, hyperthermia)
* History of cardiac disease including coronary artery disease (CAD) and cardiac dysrhythmia
* History of stroke
* History of seizure disorder
* ESRD
* Prison patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA physical status 1-3 subjects with cocaine use disorder who are scheduled to undergo surgery.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-04; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Adverse intraoperative cardiovascular events | Intraoperatively, from the time of "anesthesia start" until "anesthesia end," generally 2-4 hours
  Proportion of total anesthesia duration that mean arterial pressure (MAP) <65 or >105
Adverse postoperative cardiovascular events | Postoperatively up to 24 hours
  Increase in the postoperative troponin value compared to the patient¹s baseline preoperative troponin value

SECONDARY OUTCOMES:
The percentage of volatile anesthetic used | Intraoperatively, from the time of "anesthesia start" until "anesthesia end," generally 2-4 hours
  Average minimum alveolar concentration sevoflurane

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon TS, Pak TJ, Kim A, Gonzales MX, Volnov Y, Wright E, Vu KQ, Lu RD, Sharifi A, Minhajuddin A, Chen JL, Fox PE, Gasanova I, Fox AA, Stewart J, Ogunnaike B. A Positive Cocaine Urine Toxicology Test and the Effect on Intraoperative Hemodynamics Under General Anesthesia. Anesth Analg. 2021 Feb 1;132(2):308-316. doi: 10.1213/ANE.0000000000004808. PMID 32304462